CLINICAL TRIAL: NCT03743454
Title: Relationship Between Physical Activity Level And Physical Activity Awareness In Young Adults
Brief Title: Physical Activity Level and Physical Activity Awareness
Status: Completed | Type: Observational
Sponsor: Trakya University (Other)
Responsible Party: Principal Investigator, Nimet Sermenli Aydın, Research Assistant, Trakya University
Other Study IDs: TUTF-BAEK 2018-159
Record Dates: First submitted 2018-11-13; First posted 2018-11-16 (Actual); Last update posted 2019-01-30 (Actual); Status verified 2019-01

CONDITIONS: Physical Activity; Awareness
Keywords: physical activity level; physical activity awareness
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Men
  Interventions: Other: No intervention
- Women
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention will be applied.

SUMMARY:
It is important to determine the attitudes and behaviors of individuals towards regular exercise participation in order to direct individuals to physical activity or to implement effective practices related to increasing their participation.

The aim of this study was to determine the awareness of physical activity in young adults, the relationship between physical activity awareness and physical activity level and to investigate the differences between sexes.

ELIGIBILITY:
Inclusion Criteria:

* healthy young females and males who want to participate to the study
* individuals who have smartphones

Exclusion Criteria:

* have orthopedic, physiologic, psychiatric, neurologic or systemic disorders
* have present medication

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Study Population: healthy volunteers
Sampling Method: Non-Probability Sample
Enrollment: 403 (Actual)
Dates: Start 2018-11-21 (Actual); Primary Completion 2018-12-01 (Actual); Study Completion 2019-01-01 (Actual)

PRIMARY OUTCOMES:
Physical Activity Level | After the individuals permission, its taken in the first minute.
  Physical activity will be assessed with IPAQ-SF questionnaire. IPAQ-SF is a self-report questionnaire that assesses PA in the last 7 days. Using the IPAQ-SF scoring system, the total number of days and minutes of PA were calculated for each participant as recommended in the IPAQ website. The IPAQ-SF records the activity in four intensity levels: sitting, walking, moderate intensity (e.g., leisure cycling), and vigorous intensity (e.g, running or aerobics).
Physical Activity Awareness | After they completed the IPAQ-SF, its taken in the sixth minute.
  Physical activity awareness will be assessed with Cognitive Behavioral Physical Activity Questionnaire (CBPAQ). The CBPAQ scale consists of 15 items, including three sub-dimensions: personal barriers, outcome expectations and self-regulation. The individual items are rated at 1-5 according to the situation in which they are most appropriate. The higher the score, the higher the level of awareness.

SECONDARY OUTCOMES:
Number of Steps | After the individuals permission, number of steps will be taken at the end of the first week.
  Number of steps will be evaluated by smartphone pedometer. Pedometer provides data about the number of steps taken by the individual, so it accurately measures the individual's walking activity only. Individuals which has less than 5000 steps per day were classified as "sedentary", 5000-7499 steps "low active," 7500-9999 "somewhat active" and 10000 steps and more were classified as 'active'. Number of steps per week will be taken from individuals and mean steps per day will be calculated from number of steps per week.

CONTACTS AND LOCATIONS:
Locations (1):
- Nimet Sermenli Aydın, Edirne, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided